CLINICAL TRIAL: NCT00249756
Title: Re-Entry MTC for Offenders With MICA Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-19982-1; R01DA019982 (NIH); R01-19982-1
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Mental Disorders; Substance-Related Disorders
Keywords: Criminal Justice
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Re-entry Modified Therapeutic Community (Re-entry MTC) (Experimental)
  Interventions: Behavioral: Re-entry Modified Therapeutic Community (Re-entry MTC)
- Parole Supervision and Case Management (Active Comparator)
  Interventions: Behavioral: Parole Supervision and Case Management

INTERVENTIONS:
Behavioral: Re-entry Modified Therapeutic Community (Re-entry MTC) — In general, the MTC program model applies three fundamental adjustments - increased flexibility, decreased intensity, and greater individualization. The central TC feature is retained; the MTC, like all TC programs, seeks to develop a subculture where clients learn through self-help and affiliation with the community to foster change in themselves and others. From this base (as elaborated below), further adaptations for the population of offenders with MICA disorders were incorporated to include an emphasis on modifying criminal thinking and behavior; on recognizing and responding to the interrelationship of substance abuse, mental illness, and criminality (triple recovery); and on using strategies for symptom management.
  Arms: Re-entry Modified Therapeutic Community (Re-entry MTC)
Behavioral: Parole Supervision and Case Management — Recognizing the complexity of issues facing offenders returning to the community, and the importance of continuity of care, the CDOC established a system of aftercare substance abuse services for offenders on parole or placed in Community Corrections facilities. The statewide treatment options for the offenders consist of a network of community-based clinics and halfway houses throughout Colorado that provide substance abuse services and mental health services. Parole officers and Community Corrections case managers monitor treatment compliance to support participation in prescribed services.
  Arms: Parole Supervision and Case Management

SUMMARY:
The purpose of this study is to examine the transition of offenders with both mental illness and chemical abuse (MICA) disorders from prison to the community, where continued treatment is generally considered necessary to sustain gains made by prison treatment, and to achieve successful outcomes. The project will determine the effectiveness of a modified therapeutic community (Re-Entry MTC) approach as compared to the case management and parole supervision currently provided. The study will also assess the relative impact on treatment outcomes of the type of treatment received while in prison and of the progress achieved in re-entry treatment.

DETAILED DESCRIPTION:
Offenders having both mental illness and chemical abuse (MICA) disorders are a population of interest, in part because their special needs place exceptional demands on criminal justice and treatment systems, as well as on individuals and families. This study examines the crucial point of transition from prison to the community, where continued treatment for offenders is generally considered necessary to sustain gains made by prison treatment efforts, and to achieve successful outcomes. The project has two specific aims; Aim 1 is to test the effectiveness of Re entry MTC treatment relative to a control condition, and Aim 2 is to assess the relative impact on treatment outcomes of the type of treatment received while in prison and of the progress achieved in re-entry treatment.

On their release from prison, male offenders with MICA disorders who elect to participate in this study (N = 332), will be placed in either the experimental condition, (E) Re-entry Modified Therapeutic Community (Re-entry MTC) or the control condition, (C) Parole Supervision and Case Management currently provided, using a randomized block assignment procedure. The research employs a prospective, longitudinal, repeated measures assessment with five data collection points: baseline (Time 1, or T1) corresponding to entry into the Community Corrections facility and at 3 (T2), 6 (T3), 12 (T4), and 18 (T5) months post-baseline. The major study hypothesis is that the E condition (compared to the C condition) will produce significantly greater improvement in the presenting problems of the study participants, as measured by substance use, mental health symptoms, and criminal activities.

This project will advance scientific knowledge through a controlled study of the effectiveness of the MTC model, with demonstrated success in community settings, as a re-entry strategy for offenders with MICA disorders, thereby expanding the range of treatment models available to such clients in the community. In addition, the study will examine the degree to which prior prison treatment moderates the effectiveness of the Re-entry MTC, or the extent to which positive outcomes are independent of the type of treatment received during the prior incarceration. This distinction will inform program planning by establishing the value of MTC treatment in prison plus MTC during re-entry versus MTC re-entry treatment alone. Finally, the study tests a specific hypothesis about the degree to which the effectiveness of Re-entry MTC treatment is mediated by client progress during reentry, which will increase our understanding of the relationship between progress in treatment and post-treatment outcomes for offenders with MICA disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male offenders with serious mental illness and co-occurring chemical abuse (MICA) disorders, as the term is currently applied in the CDOC Chemical abuse consists of any substance use or dependence disorder[s] diagnosis. Serious mental disorder[s] diagnosis includes DSM IV categories for: Bipolar Mood Disorders; Major Depressive Disorder; Paranoid/Delusional Disorders; Schizophrenic Disorders; Schizoaffective Disorder; and Post Traumatic Stress Disorder.

Exclusion Criteria:

* The study has no exclusion criteria other than programmatic criteria that exclude offenders who constitute a threat to themselves or to others in the community, as determined by the Community Corrections Board at the time the offender is placed in a Community Corrections facility.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Actual)
Dates: Start 2005-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
CTCR Baseline & Follow-Up Protocol (CTCR Protocol) | Baseline and at 3, 6, 12, and 18 months
  The CTCR Protocol (CTCR, 1992) is a structured interview adapted from the ASI and DATAR for use in community treatment and the criminal justice system. The CTCR Protocol assesses these domains: socio-demographic background, substance use, psychosocial functioning, criminal justice involvement, education, employment, parenting, peer and family relations, and health. Measures of independent living skills and community functioning will be added.
Colorado Department of Corrections Record Information System (CDOC-RIS) | At 6, 12, and 18 months
  The CDOC-RIS will provide data on: charge on which incarceration is based; previous charges; current sentence; status of violent offenses; urine toxicological information on drug and alcohol use; medical information; dates of prior incarcerations; disciplinary reports; all services received while in prison; offenses committed post-release, reincarcerations, parole information (including entry into substance abuse treatment).
  Taking appropriate steps to protect inmate confidentiality, study staff will obtain the basic digital records data (and appropriate updates).
Biological Specimens | At 12 and 18 months
  Samples for urine toxicology tests will be collected on all subjects at T4 & T5, to corroborate self-report data and to provide a separate outcome measure. A reliable laboratory (e.g., Dominion Diagnostics) will test specimens for marijuana, cocaine, opiates, amphetamines, barbiturates, benzodiazepines, and ethanol; these tests are accurate for use in the preceding 48-72 hours.
Diagnostic Interview Survey-IV (DIS-IV) | At baseline
  The DIS-IV (Robins, Cottler, Bucholz & Compton, 1995) is a structured clinical interview to generate DSM-IV lifetime and current psychiatric and substance use/abuse diagnoses. The DIS-IV requires interviewer training, but not clinical expertise.
Beck Depression Inventory-II (BDI-II) | At baseline and 3, 6, 12, and 18 months
  The BDI-II (Beck, Steer, & Brown, 1996) measures Somatic Depression & Cognitive Depression and provides a Total Depression Score, consistent with the DSM-IV criteria for depressive disorders.
Symptom Checklist 90-R (SCL90-R) | At baseline and 3, 6, 12, and 18 months
  The SCL90-R (Derogatis, 1992) measures 9 domains, including somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, which provides a global index of distress, the Global Severity Index (GSI).
Rosenberg Self-Esteem (R-SES) | At baseline and 3, 6, 12, and 18 months
  The R-SES (Rosenberg, 1965) is the most widely used global measure of self-esteem, reflecting the MTC emphasis on building self-esteem, and provides positive measures of psychological status to augment the symptom pictures obtained by the other standardized psychological measures.
Measures of Social Network (adapted) | At baseline and 3, 6, 12, and 18 months
  The study will employ measures of social network adapted from existing sociometric studies to assess the building of a supportive community during and post re-entry treatment (e.g., Longabaugh et al., 1993; Neaigus et al., 1996; Rosenbaum, Nuttbrock & Magura, 1997) and to ask respondents about their most important social networks based on contact in the last 30 days. These measures are accompanied by available software for sociometric analysis (e.g., UCINET)
Client Assessment Inventory (CAI) & Staff Assessment Summary (SAS) | At 3 and 6 months
  The CAI and SAS (Kressel, 1998) measure client and staff perceptions of client progress and participation in TC treatment in 14 domains:
  maturity, responsibility, values, drug/criminal life style, maintaining images, work attitude, social skills, cognitive skills, emotional skills, sense of well being, accepting program structure and philosophy, participating in group activities, attachment to, and investment in, the program.
  The latter two scales provide measures of participation and commitment.
Therapeutic Community Scale of Essential Elements Questionnaire(SEEQ) | administered monthly over the first six months of the project and quarterly thereafter
  The study will use the SEEQ (Melnick & De Leon, 1999; Melnick et al., 2000) to capture the congruence between the program as implemented and the TC model, and using special MTC re-entry scales to describe the re-entry program.
Treatment Services Review (TSR) | administered monthly over the first six months of the project and quarterly thereafter
  The TSR (McLellan et al., 1989) is a self-report instrument that includes items on the number of times the subject received any of five types of specialized treatment services for psychological problems during a given time period (30 days).
Program Monitoring Form (PMF) | administered monthly over the first six months of the project and quarterly thereafter
  The PMF (Sacks, 1995) lists specific interventions and identifies three critical components for each intervention. The PMF will be adapted to assess intervention activities and components within each intervention and administered by research staff to clients in both E and C conditions.

SECONDARY OUTCOMES:
Quality of Employment Survey (QES) | At baseline and 3, 6, 12, and 18 months
  The measures of employment (duration and stability, hours worked, income, and occupational prestige) will be adapted from the 1977 QES (Quinn & Staines, 1979).
The Quality of Life Interview (QLI) - short form | At baseline and 3, 6, 12, and 18 months
  The original QLI (Lehman, Passidente & Hawker, 1986) was modified and shortened by NDRI staff. The instrument measures clients' satisfaction with aspects of their lives important to successful functioning in the community (e.g., family, social relations, finances, health).

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Sacks, Ph.D., Principal Investigator — National Development and Research Institutes, Inc.
Locations (3):
- United States (3):
  - Arrowhead Correctional Facility, Caqon City, Colorado
  - San Carlos Correctional Facility, Pueblo, Colorado
  - Sterling Correctional Facility, Sterling, Colorado

REFERENCES:
- [Derived] Sacks S, Chaple M, Sacks JY, McKendrick K, Cleland CM. Randomized trial of a reentry modified therapeutic community for offenders with co-occurring disorders: crime outcomes. J Subst Abuse Treat. 2012 Apr;42(3):247-59. doi: 10.1016/j.jsat.2011.07.011. Epub 2011 Sep 22. PMID 21943810